CLINICAL TRIAL: NCT06275958
Title: DOSAGE Study: a Multicenter Randomized Phase III Trial of DOSe-reduced Chemotherapy for Advanced Colorectal Cancer in Older Patients
Brief Title: DOSAGE Study: Upfront Dose-Reduced Chemotherapy in Older Patients with Metastatic Colorectal Cancer
Acronym: DOSAGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Colorectal Cancer Group (Other)
Responsible Party: Principal Investigator, Johanna E A Portielje, MD PhD, Professor Medical Oncology, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506115-17; 2023-506115-17 (EudraCT Number)
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Older Patients; Colorectal Cancer; Metastatic Cancer; Candidates for Palliative Chemotherapy
Keywords: Dose-reduced Chemotherapy; Upfront Reduction; Palliative Chemotherapy; Non-inferiority
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: A phase III, open-label, non-inferiority, randomized controlled clinical trial comparing dose-reduced chemotherapy versus standard dose chemotherapy in older adults with metastasized colorectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Doublet therapy, full dose (low toxicity risk based on G8) (Active Comparator): Low risk of toxicity: G8-score of 15 or higher
  Interventions: Drug: Doublet Chemotherapy, Standard Dose (100%)
- Doublet therapy, dose-reduced (low toxicity risk based on G8) (Experimental): Low risk of toxicity: G8-score of 15 or higher
  Interventions: Drug: Doublet Chemotherapy, Dose-reduced (75%)
- Fluoropyrimidine monotherapy, full dose (high toxicity risk based on G8) (Active Comparator): High risk of toxicity: G8-score of 14 or lower or judged as "high toxicity risk" by their treating oncologist
  Interventions: Drug: Monotherapy, Standard Dose (100%)
- Fluoropyrimidine monotherapy, dose-reduced (high toxicity risk based on G8) (Experimental): High risk of toxicity: G8-score of 14 or lower or judged as "high toxicity risk" by their treating oncologist
  Interventions: Drug: Monotherapy, Dose-reduced (75%)

INTERVENTIONS:
Drug: Doublet Chemotherapy, Standard Dose (100%) — Capecitabine 1000mg / m2 oral at day 1-14 (every 3 weeks) Oxaliplatin 130mg/m2 at day 1 (every 3 weeks) OR 5-FU 400mg/m2 IV bolus at day 1 followed by 2400mg/m2 in 46 hours (every 2 weeks) Leucovorin 400mg/m2 day 1 (every 2 weeks) Oxaliplatin 85mg/m2 day 1 (every 2 weeks)
  Arms: Doublet therapy, full dose (low toxicity risk based on G8)
Drug: Doublet Chemotherapy, Dose-reduced (75%) — 75% of: Capecitabine 1000mg / m2 oral at day 1-14 (every 3 weeks) Oxaliplatin 130mg/m2 at day 1 (every 3 weeks) OR 5-FU 400mg/m2 IV bolus at day 1 followed by 2400mg/m2 in 46 hours (every 2 weeks) Leucovorin 400mg/m2 day 1 (every 2 weeks) Oxaliplatin 85mg/m2 day 1 (every 2 weeks)
  Arms: Doublet therapy, dose-reduced (low toxicity risk based on G8)
Drug: Monotherapy, Standard Dose (100%) — - Capecitabine 1000mg/m2 oral at day 1-14 (every 3 weeks)
  Arms: Fluoropyrimidine monotherapy, full dose (high toxicity risk based on G8)
Drug: Monotherapy, Dose-reduced (75%) — 75% of:
  - Capecitabine 1000mg/m2 oral at day 1-14 (every 3 weeks)
  Arms: Fluoropyrimidine monotherapy, dose-reduced (high toxicity risk based on G8)

SUMMARY:
The goal of this phase III, open-label, non-inferiority randomized controlled clinical trial is compare upfront dose-reduced chemotherapy with the standard dose chemotherapy in older patients ( ≥70 years) with metastasized colorectal cancer, with regard to progression-free survival (PFS). The choice between monotherapy (a fluoropyrimidine) and doublet chemotherapy (a fluoropyrimidine with oxaliplatin) will be made for each individual patient based on expected risk of chemotherapy toxicity (according to the G8 screening). Patients classified as low risk of toxicity will be randomized between doublet chemotherapy in either full-dose, or with an upfront dose-reduction of 25%. Patients classified as high risk will be randomized between monotherapy in either full-dose or upfront dose-reduction.

Primary outcome is PFS. Secondary endpoints include grade ≥3 toxicity, QoL, physical functioning, overall survival, number of treatment cycles, dose reductions, hospital admissions, cumulative received dosage and cost-effectiveness.

DETAILED DESCRIPTION:
Treating older adults with chemotherapy remains a challenge, as they are strongly underrepresented in clinical trials and no robust guidelines for treating older patients exist. Moreover, older adults are at increased risk of chemotherapy-related toxicity, resulting in decreased quality of life (QoL), increased hospital admissions and high health care costs. Therefore, the aim of the DOSAGE study is to demonstrate that upfront dose-reduced chemotherapy in patients with metastasized colorectal cancer is non-inferior to full-dose treatment with regard to progression-free survival (PFS). Treatment plans (monotherapy or doublet chemotherapy) will be based on expected risk of treatment toxicity for the individual patient (according to the Geriatric 8 (G8) questionnaire). The investigators expect that this treatment strategy will lead to less grade ≥3 toxicity, less early treatment continuation and hospitalizations and a better QoL and physical functioning.

The DOSAGE study is a phase III, open-label, non-inferiority, randomized controlled clinical trial in patients aged ≥70 years with metastasized colorectal cancer eligible for palliative chemotherapy. All participating patients will undergo geriatric screening by the G8 questionnaire and will be classified as "low risk of toxicity" (G8-score of 15 or higher) or "high risk of toxicity" (G8-score of 14 or lower or judged as "high toxicity risk" by their treating oncologist). Patients classified as low risk will be randomized between a fluoropyrimidine and oxaliplatin in either full-dose, or with an upfront dose-reduction of 25%. Patients classified as high risk will be randomized between fluoropyrimidine monotherapy in either full-dose or upfront dose-reduction. Addition of targeted treatment (bevacizumab or epidermal growth factor receptor (EGFR) inhibition) is allowed. Patients with a moderate renal impairment (GFR 30- 50 mL/min) will be treated with 25% reduced starting dose of capecitabine when randomized for full dose treatment and treated with 40% reduced starting dose when randomized for upfront dose reduction.

Primary outcome is PFS. Secondary endpoints include grade ≥3 toxicity, QoL, physical functioning, overall survival, number of treatment cycles, dose reductions, hospital admissions, cumulative received dosage and cost-effectiveness. Given a non-inferiority margin of 8 weeks, 587 patients will be included (293/292 patients per arm).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years or older with colorectal cancer and distant metastases without localized treatment options.
* Patients who are candidates for first-line palliative chemotherapy as judged by their treating oncologist
* Being able to understand the Dutch language
* Adequate bone marrow and organ function: Absolute neutrophil count (ANC) > 1.5 x 10^9 mmol/L, Hemoglobin (Hb) > 6.0 mmol/L, Platelets >100 x 109 / L, Serum bilirubin ≤ 2 x upper limit of normal (ULN), serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases.

Exclusion Criteria:

* Patients who received prior palliative chemotherapy
* Patients in whom local treatment of metastases is scheduled (i.e. liver surgery or stereotactic radiotherapy)
* Candidates for triple chemotherapy
* Patients who received prior adjuvant chemotherapy in the one year before inclusion in the study (chemotherapy before that time is allowed)
* Patients with complete or incomplete dihydropyrimidine dehydrogenase (DPD) deficiency
* Patients with Microsatellite instable (MSI)-high colorectal cancer
* Patients with HIV or active hepatitis
* Patients with severe kidney failure (defined as GFR ≤30ml/min)
* Patients with severe cognitive deficits making informed consent not possible

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 587 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Time from randomization until either radiological or clinical progression or death, whichever occurs first, assessed up to at least one year.

SECONDARY OUTCOMES:
Quality of Life Questionnaire | At 1, 3, 6 and 12 months after randomization
  Measured by EQ-5D questionnaire
Quality of Life Questionnaire | At 1, 3, 6 and 12 months after randomization
  Measured by EORTC Core QLQ-C30 questionnaire
Physical functioning Questionnaire | At 1, 3, 6 and 12 months after randomization
  Measured by Lawton-Instrumental Activities of Daily Living (IADL) questionnaire
Physical functioning Questionnaire | At 1, 3, 6 and 12 months after randomization
  Measured by Katz-Activities of Daily Living (ADL) questionnaire
Grade 3-5 chemotherapy-related toxicity | Through study duration, an average of 8 months
  According to the CTCAE V5
Overall Survival | Time between randomization until death, assessed up to at least one year.
Number of completed treatment cycles | Through study duration, an average of 8 months
Dose reductions during treatment | Through study duration, an average of 8 months
  Defined as ≥25% reduction of the initial dosage
Dose delay during treatment | Through study duration, an average of 8 months
Unplanned hospitalizations | The first year after treatment initiation
Cumulative received dosage | Through study duration, an average of 8 months
  Adjusted for BSA
Cost-effectiveness | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Johanneke Portielje, Professor, Principal Investigator — Leiden University Medical Center; Joosje Baltussen, MD, Study Director — Leiden University Medical Center
Locations (36):
- Netherlands (36):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC, Amsterdam
  - Rijnstate, Arnhem
  - Wilhelmina Ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Treant, Emmen
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Beatrixziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Saxenburgh, Hardenberg
  - St. Jansdal Ziekenhuis, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Tergooi MC, Hilversum
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Laurentius Ziekenhuis, Roermond
  - Bravis ziekenhuis, Roosendaal
  - Ikazia Ziekenhuis, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Ommelander Ziekenhuis, Scheemda
  - ZorgSaam Zorggroep Zeeuws-Vlaanderen, Terneuzen
  - Haaglanden Medisch Centrum, The Hague
  - Hagaziekenhuis, The Hague
  - Bernhoven, Uden
  - Diakonessenhuis, Utrecht
  - St Antonius, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Streekziekenhuis Koninging Beatrix, Winterswijk
  - Zaans Medisch Centrum, Zaandam

IPD SHARING:
Plan to Share IPD: Yes
Which parts of your data(sets) will you select for publication?
  The datasets generated during and/or analysed during the study will not be publicly available due to participant privacy but will be available from the corresponding author on reasonable request
  Are there any restrictions placed on sharing/reuse of some/all of your data due to one or more of the following options? Signed informed consent Research agreement
  Will you publish your data open access or with restricted access? Restricted access
  Publishing your data (partly) with 'restricted access': what is the reason for this? Data contains privacy-sensitive information Contractual obligations Reuse by third-party through DSA.
  Where will you publish your (meta)data? I will not publish (meta)data outside the LUMC
Supporting Information: Study Protocol, ICF
Time Frame: The datasets generated and/or analysed during the current study are not publicly available due to patient privacy but are available from the corresponding author on reasonable request

REFERENCES:
- [Derived] Baltussen JC, van den Bos F, Slingerland M, Binda TRR, Liefers GJ, van den Hout WB, Fiocco M, Verschoor AJ, Cloos-van Balen M, Holterhues C, Houtsma D, Jochems A, Spierings LEAMM, van Bodegom-Vos L, Mooijaart SP, Gelderblom H, Speetjens FM, de Glas NA, Portielje JEA. DOSAGE study: protocol for a phase III non-inferiority randomised trial investigating dose-reduced chemotherapy for advanced colorectal cancer in older patients. BMJ Open. 2024 Aug 13;14(8):e089882. doi: 10.1136/bmjopen-2024-089882. PMID 39142680
- See also: DCCG Website — https://dccg.nl/trial/dosage